CLINICAL TRIAL: NCT03867071
Title: Early Administration of Recombinant Erythropoietin (RHEPO) in Transfusion Savings in Trauma Patients
Acronym: EPREX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PHRCI/2004/AC-01
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erythropoietin (EPO) group (Experimental)
  Interventions: Other: recombinant erythropoietin injection
- Placebo (PLA) group (Placebo Comparator)
  Interventions: Other: placebo injection

INTERVENTIONS:
Other: recombinant erythropoietin injection — Intravenous injection of 300 international units (IU) per kg (kg) of recombinant erythropoietin with a maximum of 20.000 IU, daily for a maximum of 10 days (D0 to D9).
  Arms: erythropoietin (EPO) group
Other: placebo injection — Intravenous injection 0,9% saline solution.
  Arms: Placebo (PLA) group

SUMMARY:
The objective of our study is to demonstrate the interest of early administration of recombinant erythropoietin in trauma patients

DETAILED DESCRIPTION:
Could an early use of rHuEPO (recombinant Human ErythroPOietin ) be lead to an individual benefice on transfusion savings after traumatic surgery?

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 65 years old
* Patient with an ASA 1 or 2 (ASA 1 corresponding to a patient in perfect health and ASA 2 to a patient with moderate involvement and well controlled organ function)
* patient presenting at least one of the following fractures: Basin and / or femur with surgical indication, associated or not with other fractures.
* patient with hemoglobin between 9 and 13 g / dl at the time of admission on trauma department

Exclusion Criteria:

* patient with contraindication to synthetic erythropoietin
* Patient with intravenous iron contraindication
* pregnant patient or with a risk of pregnancy
* patient who has not given his consent or does not understand the protocol
* Patient with hemodynamic instability
* patient participating in another research protocol for less than 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
number of administered red blood cells | Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Nimes university hospital, Nîmes, France